CLINICAL TRIAL: NCT04014374
Title: Post-authorization Safety Study of Allogeneic Hematopoietic Stem Cell Transplantation in Patients Treated With Mogamulizumab
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: SC18-09
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Leukemia/Lymphoma; Cutaneous T Cell Lymphoma; ATLL
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia-Lymphoma, Adult T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transplant Arm: Patients with CTCL or ATLL who received mogamulizumab within one year prior or up to 18 months after alloHCT
- Control Arm: Patients who have undergone alloHCT without exposure to mogamulizumab pre- or post-alloHCT

SUMMARY:
This is a non-interventional cohort study evaluating non-relapse mortality and toxicities in patients with CTCL or ATLL treated with mogamulizumab pre- or post- alloHCT for patients transplanted beginning January 1, 2012 until accrual is complete.

DETAILED DESCRIPTION:
This is an observational, retrospective and prospective study where subjects who have received mogamulizumab either within one year before or within 18 months after transplantation will be followed for data collection. Data will be collected at baseline (retrospectively), 100 days post alloHCT, 6-months, 1 year and at 2 years post alloHCT (retrospectively and prospectively).

A cut-off time limit of 18 months post alloHCT exposure will allow at least 6 months of follow-up within the 2 years post-alloHCT follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered to the Center for International Blood and Marrow Transplant Research (CIBMTR)
* Adults ≥18 years of age with either CTCL or ATLL;
* AlloHCT performed from January 2012 onward.

Exclusion Criteria:

• Patients without consent for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include a minimum of 50 patients with CTCL or ATLL who received mogamulizumab within one year prior to alloHCT. At least 40 patients should have been diagnosed with CTCL and at least 33 patients should have received mogamulizumab as last therapy line before alloHCT. Data will be collected from no more than 100 controls with similar characteristics to the mogamulizumab-treated patients, and who have undergone alloHCT without exposure to mogamulizumab pre- or post-alloHCT. Information on patients receiving mogamulizumab within 18 months after alloHCT will also be collected.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Assess toxicities or complications of transplant among patients who were treated with mogamulizumab, alone or in combination | one year prior to alloHCT to within 18 months after alloHCT
  This study will utilize comprehensive report form (CRF) data, modified transplant essential data (TED) and supplemental data. In patients with only TED data the supplemental data will provide the required additional information for data analyses to meet the objectives of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CIBMTR, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No